CLINICAL TRIAL: NCT06688227
Title: Effects Of Isolated And Integrated Core Stability Training On Power, Balance And Performance In Fast Bowlers
Brief Title: Effects Of Isolated And Integrated Core Stability Training In Fast Bowlers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0425
Record Dates: First submitted 2024-10-17; First posted 2024-11-14 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Core Strength; Power; Balance
Keywords: Core Strenght; Power; Balance; core stability; Integrated Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isolated Core Stability Program (Other): The control group consists of basic core exercises which include the activation of transversusabdominins and multifidus muscles and progressive strengethening of these muscles in all positions using swiss balls and floor mats. All exercises were done for at least 3 sets of 15 repetitions to build proper core stability.
  Interventions: Other: Isolated Core Stability Program
- Integrated Core Stability Program (Experimental): An individualized protocol was designed for these cricketers targeting static and dynamic core stability, with integration of balance, endurance and power component.
  Tranversusabdominis and multifidus strengthening is combined with upper extremity motions to work on the fast bowling action i.e throwing of the players.
  At the same time lower extremity balance and strengthening is also included to ensure the high speed of sprint.
  Interventions: Other: Integrated Core Stability Program

INTERVENTIONS:
Other: Isolated Core Stability Program — The control group consists of basic core exercises which include the activation of transversusabdominins and multifidus muscles and progressive strengethening of these muscles in all positions using swiss balls and floor mats. All exercises were done for at least 3 sets of 15 repetitions to build proper core stability.
  Arms: Isolated Core Stability Program
Other: Integrated Core Stability Program — An individualized protocol was designed for these cricketers targeting static and dynamic core stability, with integration of balance, endurance and power component.
  Tranversusabdominis and multifidus strengthening is combined with upper extremity motions to work on the fast bowling action i.e throwing of the players.
  At the same time lower extremity balance and strengthening is also included to ensure the high speed of sprint.
  Arms: Integrated Core Stability Program

SUMMARY:
The objective of this study will be to compare the effects of isolated and integrated core stability training on power, balance and performance in fast bowlers.

DETAILED DESCRIPTION:
Athletes consistently strive for improved performance, often incorporating strength and conditioning routines that inevitably include elements of core strengthening. The crucial question emerges: how does enhancing core strength and stability contribute to elevated athletic performance? Before delving into this issue, it is essential to clarify the concept of core strength and stability. The core consists of both passive and active components, including bones, muscles, and ligaments in the lumbar spine, pelvis, and hips. Core strength is characterized by the capacity of the core muscles to produce and sustain force. In contrast, core stability emphasizes the significance of passive and active stabilizing elements within the lumbo-pelvic area. Beyond mere strength, core stability denotes the adeptness of these stabilizers to uphold proper trunk and hip posture, equilibrium, and control during both stationary and kinetic activities. It can be conceptualized as the ability to sustain command over the core while exerting core strength or when met with external disruptions.

The objective of this study will be to compare the effects of isolated and integrated core stability training on power, balance and performance in fast bowlers. This study will be a Randomized Clinical trial. Data will be collected fromPakistan Sports Board, Lahore. Subjects fulfilling the inclusion criteria will be included in this study. Baseline measurements will be taken before the application of interventions. Treatment will be then given to control and intervention group according to their allocation. Post-Treatment values for the baseline measures will be taken. Pre, 6th week and 12th week post treatment values will be analyzed. All subjects received a total of three treatment sessions in a week over the period of 12 weeks. The data will be analyzed using SPSS v 25.

ELIGIBILITY:
Inclusion Criteria:

* • Age group: 18 to 28 years. Individuals younger than 18 needed parental consent, and those older than 30 faced a higher likelihood of degeneration in the thoracic and lumbar spine region

  * No history of lower back pain
  * Gender: Male. Considering the differences in anatomy and physiology between males and females, it was deemed advantageous to concentrate solely on one gender to ensure continued homogeneity
  * They had actively participated in Action Cricket within one of the intermediate leagues for a minimum of six months

Exclusion Criteria:

* Athletes with physical disability and major health problems.
* Not willing to participate.
* Patients with MSK disorders.
* Female athletes will not be included because of anatomical and physiological differences.
* Participants with a recent history of significant injuries, especially those related to the core or lower extremities, as this could confound the study results.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Seated Medicine Ball Throw Test (SMBT): | 12 weeks
  The seated medicine ball throw (SMBT) serves as a field test designed to evaluate upper-body muscular power by gauging the maximum distance an individual can propel a medicine ball from a seated position. This assessment is cost-effective and easier to integrate into a field test battery compared to alternative methods for evaluating upper body power. Demonstrating validity and reliability, participants engage in the SMBT by throwing a 2 kg medicine ball with a 19.5 cm diameter while positioned on the floor, with the upper torso against the wall and legs extended, maintaining a trunk angle of 90°.
Sit Up Test (SUT) | 12 weeks
  The participant assumes a supine position on the floor, with knees flexed at a 90° angle, hands positioned beside their head, and elbows directed straight forward. A proper execution of the sit-up involved touching the elbows to the knees and then returning to the starting position, ensuring that the shoulders made contact with the floor. The number of repetitions completed was documented to quantify the level of endurance achieved in each trial. Exhaustion, defined as the inability to execute another repetition, marked the conclusion of the test. The Sit-Up Test (SUT), characterized by its simplicity of administration and low costs, proved to be an effective tool for assessing muscle endurance
Star Excursion Balance Test (SEBT): | 12 weeks
  The SEBT was initially outlined with the individual positioned at the center of eight lines forming an eight-pointed star, each with a 45° separation. Subsequent studies demonstrated that this approach could be streamlined with just three lines, referred to as anterior (ANT), posteromedial (PM), and posterolateral (PL), based on the stance foot. This simplified version, commonly known in the literature as the mSEBT, is now frequently employed, though not consistently. The adoption of the mSEBT helps save testing time by eliminating redundant testing directions while upholding the consistency and reliability observed in the original SEBT. Typically, the average of the three directions is calculated to generate a composite score (COMP)

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larwa J, Stoy C, Chafetz RS, Boniello M, Franklin C. Stiff Landings, Core Stability, and Dynamic Knee Valgus: A Systematic Review on Documented Anterior Cruciate Ligament Ruptures in Male and Female Athletes. Int J Environ Res Public Health. 2021 Apr 6;18(7):3826. doi: 10.3390/ijerph18073826. PMID 33917488
- [Background] Kim B, Yim J. Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial. Tohoku J Exp Med. 2020 Jul;251(3):193-206. doi: 10.1620/tjem.251.193. PMID 32669487
- See also: Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/32669487
- See also: Stiff Landings, Core Stability, and Dynamic Knee Valgus: A Systematic Review on Documented Anterior Cruciate Ligament Ruptures in Male and Female Athletes — https://pubmed.ncbi.nlm.nih.gov/33917488